CLINICAL TRIAL: NCT03553251
Title: Oral Beta-lactam Drug Reintroduction Protocol, Without Previous Skin Tests, in Children Under 16 Years of Age With a Clinical History That is Not Suggestive of Immunoglobulin E (IgE)-Mediated Anaphylaxis or Toxidermia to Beta-lactams.
Brief Title: Protocol of Reintroduction of Beta-lactams in Children at Low Risk of Anaphylaxis.
Acronym: TRO-b-lact
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC18_0193
Record Dates: First submitted 2018-05-25; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Hypersensitivity; Beta Lactam Adverse Reaction
Keywords: Hypersensitivity; Beta Lactam Adverse Reaction
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to establish the rationale for the practice of performing an oral reintroduction test without previous skin tests in children at low risk of IgE-mediated reaction or drug-induced toxidermia, and to confirm the criteria for a drug reintroduction test could be performed without previous skin tests, without subsequent risk of reaction for the child. The primary endpoint will be the risk of a severe IgE-mediated or delayed hypersensitivity reaction in children who received beta-lactam drug reintroduction protocol prior to skin testing.

ELIGIBILITY:
Inclusion Criteria:

* Children under 16 years of age coming for a consultation for a beta-lactam oral reintroduction test.

Exclusion Criteria:

* Refusal of the legal representatives of the subject for their child to participate in the study,
* If his age permits, refusal of the subject to participate in the study,
* Subject aged over 16,
* Pregnancy,
* Absence of affiliation of the subject to a social security scheme,
* Skin tests with incriminated beta-lactam already made before the consultation,
* Existence of contraindications to the realization of oral reintroduction drug test with the suspected antibiotic,
* Existence of criteria in the initial reaction suggestive of a non-low risk of IgE-mediated or delayed hypersensitivity to the incriminated beta-lactam, Taking antihistamine, corticosteroids or beta-blockers within 5 days prior to the oral reintroduction drug test,
* Travel abroad of the child scheduled within 7 days of the oral reintroduction drug test.

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children under 16 years of age with a clinical history that is not suggestive of IgE-mediated anaphylaxis or toxiderma to beta-lactams.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07-30 (Estimated); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
low risk of 2% IgE-mediated or severe delayed hypersensitivity reactions following an oral beta-lactam drug reintroduction | At the end of the study, after 2 years.
  Demonstrate a low risk of 2% IgE-mediated or severe delayed hypersensitivity reactions following an oral beta-lactam drug reintroduction, without previous skin tests, in children selected by a questionnaire as being at low risk of IgE-mediated or delayed

SECONDARY OUTCOMES:
Risk evaluation | At the end of the study, after 2 years.
  Evaluate a risk of IgE-mediated or delayed non-severe hypersensitivity reactions.
explain the occurrence of a reaction of IgE-mediated or delayed hypersensitivity | At the end of the study, after 2 years.
  If an IgE-mediated or delayed hypersensitivity reaction (s), severe or not, occurs during the oral beta-lactam drug reintroductions, analyze all the information collected in the inclusion questionnaire (s) of the patient (s) concerned, in order to find the element (s) most likely to explain the occurrence of a reaction of IgE-mediated or delayed hypersensitivity despite initial selection of patients at low risk of reaction.